CLINICAL TRIAL: NCT02520076
Title: Improving Single Donor Success Rate in Clinical Islet Transplantation Using Alpha-1 Antitrypsin (Aralast NP)
Brief Title: Aralast NP in Islet Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00047923
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Islet Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AAT treated group (Experimental): Study subjects will receive Alpha-1 Antitrypsin (AAT) study drug intravenously in 4 doses over 15 days around the time of their transplant. The islets will also be prepared in a solution of AAT.
  Interventions: Drug: Alpha-1 Antitrypsin

INTERVENTIONS:
Drug: Alpha-1 Antitrypsin — Subjects will receive their islets treated with Aralast NP during islet isolation process.
  Subjects will receive Aralast NP at a dose of 120 mg/kg (at an infusion rate of 0.2 mL/kg/min or less), dependent on patient tolerance, based on Day -1 admission weight and dose rounded to the nearest 20 mg) at the following time points:
  * Pre-transplant Day -1
  * Post-transplant Day 3
  * Post-transplant Day 7
  * Post-transplant Day 14

SUMMARY:
Islet transplantation is a relatively new procedure used in people with difficult to control Type 1 diabetes. Insulin producing cells (islets) are isolated from a pancreas donated by the next of kin of a person who is brain dead. After the cells are prepared, the islets are transplanted into the recipient's liver and produce insulin. Patients who receive an islet transplant take medication that suppresses their immune system and prevent rejection of the islet tissue.

The investigators have also learned that there is general inflammation at the time of the transplant that is not fully controlled with our standard medications. The investigators believe this inflammation may cause some islet cell death around the time of transplant. Due to this islet death around the time of transplant, most recipients need 2 or 3 separate transplant procedures.

The investigators are studying the use of Alpha-1 Antitrypsin (AAT) in islet transplant to decrease the amount of cell death caused by general inflammation. In this study, the investigators hope to decrease the need for more than one transplant procedure by controlling inflammation, before and after transplant, with Alpha-1 Antitrypsin (Aralast NP).

Alpha-1 Antitrypsin is a protein made in healthy humans that helps to prevent tissue damage during times of inflammation. Alpha-1 Antitrypsin is obtained from healthy plasma donors. There have been studies in Islet Transplant in monkeys using this medication and it has shown to protect the islets from inflammation.

This study involves using Alpha-1 Antitrypsin in addition to our current Standard of Care medications used in Islet Transplant.

DETAILED DESCRIPTION:
METHODS & PROCEDURES:

This clinical trial will be a non-randomized, open-label, single arm, prospective trial to asses the efficacy of AAT in preventing non-immunologic loss of transplanted islet mass in a single-donor islet transplant. Enrolled patients (n=12) will participate in the study for 1 year, with outcomes assessed during islet isolation, 90 days post-transplant and at 1 year post-transplant.

The current Standard of Care treatment for Islet Transplant includes induction (Alemtuzumab/Basiliximab) and long-term immunosuppression (Prograf/Cellcept). The engraftment regimen includes anti-inflammatory medications (Etanercept/Anakinra) and intravenous insulin and heparin. We will utilize the current Islet Standard of Care Protocol. The only additional intervention used in this pilot trial is the addition of the investigational agent, alpha-1-antitrypsin to islet processing, culture, and patient treatment pre- and post-transplant.

Islet Dosage and Culture

Islets will be treated with AAT (to a final dilution of 0.5mg/mL) throughout the isolation and culture process. Islet treatment will include:

* Flushing through the superior mesenteric artery and splenic artery (final dilution 0.5mg/mL)
* Culturing with AAT (final dilution 0.5mg/mL)

Participant Dosing

Subjects undergoing intraportal clinical islet transplantation will receive treatment (AAT at 120mg/kg intravenously, based on Day -1 admission weight and rounded to the nearest 20mg) at the following time points:

* Day -1 prior to transplant
* Day 3 post-transplant
* Day 7 post-transplant
* Day 14 post-transplant Recipient management including the transplant procedure, postoperative care, immunosuppression and other medications, and post-transplant monitoring will follow standard of care protocols.

SCOPE & DURATION:

Recruitment will take place at the Clinical Islet Transplant Program at the University of Alberta Hospital, Edmonton, Alberta. Participants (N=12) will be adult patients, assessed and deemed appropriate to activate on the waiting list for islet transplantation. Anticipated duration of enrollment is 12 months, with follow-up at 90 days and 12 months.

In this pilot study control data will be obtained from a Standard of Care control cohort as comparison.

We will also obtain 2 year and 3 year long-term follow-up data from standard of care testing. This long-term follow up will review data collected within 3 years post-transplant and will include the following: patient and graft survival data, biochemical data from routine blood work, routine and for cause imaging, metabolic testing, initiation of interventions to treat complications, and reporting of any adverse or serious adverse events.

STUDY FOLLOWUP:

As follow-up, this study will use a number of blood tests and parameters used by the clinical program. We will obtain the following information regarding participant outcomes from routine blood testing, metabolic testing, and clinic visits:

* Complete blood count (CBC)-differential to monitor white and red blood cells
* Liver function tests
* Kidney function tests
* Blood sugar tests, including the Hemoglobin A1c (HbA1c) which estimates average blood sugars over 3 months.
* C-peptide testing, a chemical produced only be healthy, working islets.

These clinics will occur weekly x 4weeks, then at 1 month, 3 months, 6, months and 12 months. Participants will then have annual clinic visits, all as standard of care. Clinic visits include vital signs, physician assessment, review of recorded blood glucose records, and determination of patient requiring insulin or becoming insulin independent by a set of criteria based on the above blood sugar testing and glucose records.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible the participant must have had Type 1 Diabetes Mellitus (T1DM) for more than 5 years, complicated by at least 1 of the following situations that persist despite intensive insulin management efforts:

  1. Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels < 3.0 mmol/L, indicated by, 1 or more episodes of severe hypoglycemia requiring third party assistance within 12 months, a Clarke score ≥4, HYPO score ≥1,000, lability index (LI) ≥400 or combined HYPO/LI >400/>300.
  2. Metabolic instability, characterized by erratic blood glucose levels that interfere with daily activities and or 1 or more hospital visits for diabetic ketoacidosis over the last 12 months.
* Participants must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

1. Hypersensitivity to Aralast NP, history of immunoglobulin A (IgA) deficiency, or assessed low IgA (< 0.70 g/L).
2. Severe co-existing cardiac disease, characterized by any one of these conditions: (a) recent (within the past 6months) myocardial infarction; (b) left ventricular ejection fraction <30%; or (c) evidence of ischemia on functional cardiac exam.
3. Active alcohol or substance abuse, to include cigarette smoking (must be abstinent for 6 months prior to listing for transplant).
4. Psychiatric disorder making the subject not a suitable candidate for transplantation, (e.g., schizophrenia, bipolar disorder, or major depression that is unstable or uncontrolled on current medication).
5. History of non-adherence to prescribed regimens.
6. Active infection including Hepatitis C, Hepatitis B, HIV, or tuberculosis (TB) (subjects with a positive purified protein derivative (PPD) performed within one year of enrollment, and no history of adequate chemoprophylaxis).
7. Any history of, or current malignancies except squamous or basal skin cancer.
8. BMI > 35 kg/m2 at screening visit.
9. Age less than 18 or greater than 68 years.
10. Measured glomerular filtration rate <60 mL/min/1.73 m2.
11. Presence or history of macroalbuminuria (>300 mg/g creatinine).
12. Clinical suspicion of nephritic (hematuria, active urinary sediment) or rapidly progressing renal impairment (e.g. Increase in serum creatinine of 25% within the last 3-6 months).
13. Baseline Hb < 105 g/L in women, or < 120 g/L in men.
14. Baseline screening liver function tests (LFT) outside of normal range, with the exception of uncomplicated Gilbert's Syndrome. An initial LFT panel with any values >1.5 times the upper limit of normal (ULN) will exclude a patient without a re-test; a re-test for any values between ULN and 1.5 times ULN should be made, and if the values remain elevated above normal limits, the patient will be excluded.
15. Untreated proliferative retinopathy.
16. Positive pregnancy test, intent for future pregnancy or male subjects' intent to procreate, failure to follow effective contraceptive measures, or presently breast-feeding.
17. Previous transplant or evidence of significant sensitization on panel reactive antibody (PRA) (at the discretion of the investigator).
18. Insulin requirement >1.0 U/kg/day
19. Hemoglobin A1c (HbA1c) >12%.
20. Uncontrolled hyperlipidemia [fasting LDL cholesterol > 3.4 mmol/L, treated or untreated; and/or fasting triglycerides > 2.3 mmol/L)].
21. Under treatment for a medical condition requiring chronic use of steroids.
22. Use of coumadin or other anticoagulant therapy (except aspirin) or subject with prothrombin time / international normalized ratio (PT/INR) > 1.5.
23. Untreated Celiac disease.
24. Patients with Graves disease will be excluded unless previously adequately treated with radioiodine ablative therapy.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-08; Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
To demonstrate AAT efficacy in preventing non-immunologic loss of transplanted islet mass in a single-donor islet transplant. | Day 90 post-transplant
  Insulin independence at day 90 post-transplant (initial, single-donor transplant)

SECONDARY OUTCOMES:
To demonstrate safety of AAT during islet isolation and culture | Day -1 pre-transplant
  Post-isolation measurements, compared to current standard protocol isolation data, for the following parameters:
  * Endotoxin level
  * Microbiological culture [bacterial (both aerobic and anaerobic), fungal, mycoplasma, and mycobacterium culture]
To demonstrate efficacy of AAT to improve islet isolation quantity and quality | Day -1 pre-transplant
  Post-isolation measurements, compared to current standard protocol isolation data, for the following parameters:
  * Islet yield
  * Viability (SytoGreen/ethidium bromide)
  * Purity
  * Beta cell specific viability
  * Cell composition assay
  * Glucose stimulated insulin release
  * DNA content
To demonstrate safety of AAT in islet transplantation. | Year 1 post-transplant
  Adverse Event/Serious Adverse Event morbidity within 1 year post-transplant, which includes the following:
  * Primary non-function (PNF)
  * End-organ dysfunction
  * Malignancy
  * Opportunistic infection
  * Inpatient hospitalization
  * Prolongation of existing hospitalization
  * A life-threatening event
  * Persistent or significant disability
  * Congenital anomaly or birth defect
  * Patient death
To demonstrate AAT efficacy in the prevention of long-term metabolic burn-out. | Year 1 post-transplant
  * Full graft function at 1 year after initial single-donor transplant, compared to retrospective controls (current standard of care induction).
  * Partial graft function at 1 year after initial single-donor transplant compared to retrospective controls (current standard of care induction).

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada